CLINICAL TRIAL: NCT03394807
Title: Laparoscopic Guided Regional Analgesia (LaGRA) Reduces Post Operative Pain After Laparoscopic Cholecystectomy - a Randomised, Controlled Trial.
Brief Title: LaGRA Trial in Laparoscopic Cholecystectomy
Acronym: LaGRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Health Service Executive, Ireland (Other)
Responsible Party: Principal Investigator, Des Toomey, Consultant Surgeon, Health Service Executive, Ireland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LaGRA-MRHM
Record Dates: First submitted 2017-12-15; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Regional Anesthesia Morbidity; Gallbladder Stone; Pain
MeSH Terms: conditions — Cholecystolithiasis; Pain | interventions — Levobupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LaGRA (Experimental): regional anaesthesia of the right upper quadrant by injection of levobupivacaine 0.25% to the transversus abdominis plane and the rectus sheath under laparoscopic guidance immediately following specimen removal
  Interventions: Drug: Levobupivacaine
- Placebo (Placebo Comparator): Sham regional anaesthesia of the right upper quadrant by injection of Saline 0.9% to the transversus abdominis plane and the rectus sheath under laparoscopic guidance immediately following specimen removal
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levobupivacaine — Levobupivacaine injection to Transversus abdominis plane and rectus sheath
  Other Names: Chirocaine
  Arms: LaGRA
Drug: Placebo — Saline injection to Transversus abdominis plane and rectus sheath
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This study investigated the effectiveness of a surgeon administered, laparoscopic guided, regional anaesthesia technique.

DETAILED DESCRIPTION:
A prospective, double blind, randomised controlled trial was performed. Consenting patients undergoing laparoscopic cholecystectomy were randomised, by envelope, to a laparoscopic guided 2-point blockade (subcostal transversus abdominis plane and rectus sheath) using either Chirocaine® 2.5mg/ml (LaGRA) or 0.9% Saline (Placebo) after specimen extraction.

Primary endpoints were post-operative pain in the first 6 hours. Secondary endpoints were analgesic/anti-emetic usage and day case and re-admission rates. Data was analysed using GraphPad Prism (V7).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy
* ASA I, II or III

Exclusion Criteria:

* Patients that don't consent to be included
* Allergy to levobupivacaine

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Post operative pain score | 6 hours post operatively
  Visual analogue pain scores ranging from 0 to 10

SECONDARY OUTCOMES:
Opioid use | Perioperative period including first 6 hours post operatively
  Amount (mg) of opioid medication administered
Analgesic use | Perioperative period including first 6 hours post operatively
  Type and dose of all non opioid analgesic medications prescribed
Readmission rate | 30 days post operative
  Patient readmitted to hospital for any reason
Daycase rates | Day of surgery
  Patient that was planned for daycase but admitted overnight

IPD SHARING:
Plan to Share IPD: No